CLINICAL TRIAL: NCT06287008
Title: A Comparative Study on Outcomes of ABO-Incompatible Kidney Transplants Between Robot-Assisted vs. Open Surgery: A Retrospective Cohort Study
Brief Title: ABO-Incompatible Kidney Transplants Between Robot-Assisted vs. Open Surgery
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sei Won Lee, Clinical Professor, Asan Medical Center
Other Study IDs: 2023-0085
Record Dates: First submitted 2024-02-24; First posted 2024-02-29 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Kidney Transplantation
Keywords: robot-assisted kidney transplantation; ABO incompatible; biopsy-proven acute rejection; immunologically high-risk patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum (5cc~10cc)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OKT: patients who underwent "open kidney transplantation"
- RAKT: patients who underwent "robot-assisted kidney transplantation"
  Interventions: Procedure: robot-assisted kidney transplantation

INTERVENTIONS:
Procedure: robot-assisted kidney transplantation — The interventional surgery is a robot-assisted kidney transplantation and its efficacy will be measured against that of open kidney transplantation
  Groups: RAKT

SUMMARY:
While robot-assisted kidney transplantation (RAKT) offers potential benefits such as minimal postoperative pain, better cosmesis, fewer wound infections, and shorter hospital stay, its efficacy in ABO-incompatible (ABO-i) KT compared to open KT (OKT) remains understudied. This study aims to compare ABO-i KT outcomes between RAKT and OKT.

The study utilized data from 29 ABO-i RAKT and 210 ABO-i OKT cases performed at Asan Medical Center from October 2020 to February 2023. Univariate and multivariate analyses were performed to evaluate factors associated with a composite of biopsy-proven acute rejection (BPAR), de novo donor-specific antibodies (DSA), and overall graft failure.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for living donor ABO incompatible kidney transplantation
* Presenting an IsoAgglutinin immunoglobulin G titer (anti-A-B) between 1/8 and 1/128 before operation
* Patient older than 18 years and young than 80 years
* Patient able to sign an informed consent form

Exclusion Criteria:

* Patient with comorbidities or hypersensitivity that prevent desensitization protocols
* Women who are pregnant, or who may become pregnant or breastfeeding women
* Subjects under legal protection
* Subjects participating in another interventional research protocol or in an exclusion period from another interventional research protocolPatient affiliated with a social security scheme

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: study includes 210 patients who undergo ABOi-open kidney transplantation and 29 who undergo ABOi-robot assisted kidney transplantation
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Graft survival | 1 year post-operative
  allograft (kidney) survival
renal function | 1 year post-operative
  renal function measured in terms of eGFR (Estimated Glomerular Filtration Rate)

SECONDARY OUTCOMES:
. A composite of biopsy-proven acute rejection, graft failure, and the development of de novo donor-specific antibodies | 1 year post-operative
  . A composite of biopsy-proven acute rejection, graft failure, and the development of de novo donor-specific antibodies

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim JM, Kwon HE, Ko Y, Jung JH, Kwon H, Kim YH, Shin S. A comparative study on outcomes of ABO-incompatible kidney transplants between robot-assisted vs. open surgery-propensity score-matched analysis: a retrospective cohort study. BMC Nephrol. 2024 Nov 14;25(1):410. doi: 10.1186/s12882-024-03842-1. PMID 39543527